CLINICAL TRIAL: NCT02697188
Title: Phase IIa, Pilot, Pharmacokinetic Study of Oral Testosterone Ester Formulations in Hypogonadal Men
Brief Title: Pilot Pharmacokinetic Study of Oral Testosterone Ester Formulations in Hypogonadal Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLAR-07004
Record Dates: First submitted 2014-01-29; First posted 2016-03-03 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Hypogonadism
Keywords: testosterone; male hypogonadism; low testosterone
MeSH Terms: conditions — Hypogonadism; Eunuchism | interventions — testosterone undecanoate; testosterone enanthate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Testosterone undecanoate (Experimental): Period 2 - 200 mg T (as TU) QD Period 3 - 200 mg T (as TU) BID (100 mg/dose) Period 4 - 400 mg T (as TU) BID (200 mg/dose)
  Interventions: Drug: Testosterone undecanoate
- Testosterone enanthate (Active Comparator): Period 1 - 400 mg T (as TE) QD Period 5 - 800 mg T (as TE) BID (400 mg/dose)
  Interventions: Drug: Testosterone enanthate

INTERVENTIONS:
Drug: Testosterone undecanoate — Single-day dose as QD or BID for 3 of 5 crossover periods
  Other Names: TU
  Arms: Testosterone undecanoate
Drug: Testosterone enanthate — Single-day dose for 2 of 5 crossover periods
  Other Names: TE
  Arms: Testosterone enanthate

SUMMARY:
Determine the serum pharmacokinetic profile for two oral formulations of T-esters (one TE and one TU) administered once -(QD) and twice-daily (BID) to hypogonadal men.

DETAILED DESCRIPTION:
Five period cross-over study in which subjects received a single day of dosing in each period. Dosing was either QD or BID with one of two T esters (T-enanthate (TE) or T-undecanoate (TU)). Dosing was within 5 minutes of meals (breakfast and for BID dosing dinner). There was a minimum of a 5-day washout between periods. Subjects were hypogonadal men.

ELIGIBILITY:
Inclusion Criteria:

Male, ages 18 to 65 Serum total testosterone less than or equal to 250 ng/dL Naive to androgen replacement therapy Subject must be on stable doses of thyroid or adrenal replacement hormones for at least 14 days prior to enrollment

Exclusion Criteria:

Significant intercurrent disease of any type, in particular, liver, kidney or heart disease, uncontrolled diabetes mellitus or psychiatric illness. Patients with treated hyperlipidemia will not be excluded provided they have been stable on their lipid-lowering mediation for at least three months. For non-insulin dependent diabetic subjects, HbA1c>9%.

Abnormal prostate digital rectal examination, elevated PSA (serum PSA >4ng/mL), AUA Sympton Score greater than or equal to 15 points, and a history or prostate cancer.

Serum transaminases >2X upper limit of normal (ULN) or serum bilirubin >2.0 mg/dL.

History of severe or multiple allergies, severe adverse drug reaction or leucopenia. Known hypersensitivity to lidocaine or all surgical dressings.

History of abnormal bleeding tendencies. Oral, topical, or buccal T therapy within the previous week, or intramuscular T injection within the previous 4 week.

Use of dietary supplements that may increase serum T, such as androstenedione or DHEA, within the previous 4 weeks.

Know malabsorption syndrome and/or current treatment with oral lipase inhibitors, bile acid-binding resins, colestipol, fibric acid derivatives, gemfibrozil, and probucol.

Smokers who are unable to refrain from smoking during confinement periods. History of, or current evidence of, abuse of alcohol or any drug substance. Poor compliers or those unlikely to attend. Receipt of any drug as part of a research study within 30 days of inital dose administration in this study.

Blood donation (usually 550 mL) within the 12-week period before the initial study dose.

Hematocrit less than 35%. Known clinical polycythemia or hematocrit greater than 50%. Current use of paroxetine and clomipramine, antiandrogens, estrogens, p450 enzyme inducers, or barbiturates.

History of sleep apnea.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald S Swerdloff, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center; Sherwyn Schwartz, MD, Principal Investigator — dgd Research, Inc.
Locations (2):
- United States (2):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Los Angeles, California
  - dgd Research, Inc, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cross over study with 5 periods. Twelve subjects enrolled and completed 5 crossover periods each.
Groups:
- Testosterone Enanthate and Testosterone Undecanoate: Testosterone Enanthate Periods 1 and 5 Single-day dose as QD Period 1 and BID Period 5 Testosterone Undecanoate: Single-day dose as QD Period 2 and BID Periods 3 and 4
Period: TE Period 1 - 400 mg QD
Arm/Group | Testosterone Enanthate and Testosterone Undecanoate
Started | 12
Completed | 12
Not Completed | 0
Period: TU Period 2 - 200 mg QD
Arm/Group | Testosterone Enanthate and Testosterone Undecanoate
Started | 12
Completed | 12
Not Completed | 0
Period: TU Period 3 - 200 mg BID
Arm/Group | Testosterone Enanthate and Testosterone Undecanoate
Started | 12
Completed | 12
Not Completed | 0
Period: TU Period 4 - 400 BID
Arm/Group | Testosterone Enanthate and Testosterone Undecanoate
Started | 12
Completed | 12
Not Completed | 0
Period: TE Period 5 - 800 mg BID
Arm/Group | Testosterone Enanthate and Testosterone Undecanoate
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Testosterone Enanthate and Testosterone Undecanoate: Period 1 - 400 mg T (as TE) QD Period 5 - 800 mg T (as TE) BID (400 mg/dose) Testosterone enanthate: Single-day dose for 2 of 5 crossover periods
  Period 2 - 200 mg T (as TU) QD Period 3 - 200 mg T (as TU) BID (100 mg/dose) Period 4 - 400 mg T (as TU) BID (200 mg/dose) Testosterone undecanoate: Single-day dose as QD or BID for 3 of 5 crossover periods
Arm/Group | Testosterone Enanthate and Testosterone Undecanoate
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 53 [31 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Serum Testosterone Cavg
Description: The objective of the study was to determine the single day serum pharmacokinetic profile for two oral formulations of T-esters (one TE and one TU formulation) administered once- and twice-daily to hypogonadal men.
Time Frame: Concentrations at -0.5, 0, 1, 2, 4, 8, 12, 13, 14, 16, 20, 24 and 34 hours post dose
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Enanthate and Testosterone Undecanoate
Number analyzed (Participants) | 12
ng/dL
  TE Period 1 400 mg QD | 293 (148)
  TU Period 2 200 mg QD | 246 (77)
  TU Period 3 100 mg BID | 281 (89)
  TU Period 4 200 mg BID | 385 (132)
  TE Period 5 400 mg BID | 316 (167)

2. Secondary Outcome: Mean Serum Dihydrotestosterone Cmax
Description: as for outcome 1
Time Frame: 24 hours post-dose in each period
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Enanthate and Testosterone Undecanoate
Number analyzed (Participants) | 12
ng/dL
  TE Period 1 400 mg QD | 140 (96)
  TU Period 2 200 mg QD | 122 (66)
  TU Period 3 100 mg BID | 97.9 (51.2)
  TU Period 4 200 mg BID | 114 (58)
  TE Period 5 400 mg BID | 127 (81)

ADVERSE EVENTS:
Time Frame: Subjects received doses on 5 dosing days spanning approximately 4 weeks.
Groups:
- Testosterone Enanthate 400 mg QD: Period 1: Testosterone Enanthate 400 mg QD
- Testosterone Undecanoate 200 mg QD: Period 2: Testosterone Undecanoate 200 mg QD
- Testosterone Undecanoate 100 mg BID: Period 3: Testosterone Undecanoate 100 mg BID
- Testosterone Undecanoate 200 mg BID: Period 4: Testosterone Undecanoate 200 mg BID
- Testosterone Enanthate 400 mg BID: Period 5: Testosterone Enanthate 400 mg BID
Arm/Group | Testosterone Enanthate 400 mg QD | Testosterone Undecanoate 200 mg QD | Testosterone Undecanoate 100 mg BID | Testosterone Undecanoate 200 mg BID | Testosterone Enanthate 400 mg BID
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 3/12 | 3/12 | 4/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Enanthate 400 mg QD (N=12) | Testosterone Undecanoate 200 mg QD (N=12) | Testosterone Undecanoate 100 mg BID (N=12) | Testosterone Undecanoate 200 mg BID (N=12) | Testosterone Enanthate 400 mg BID (N=12)
headache (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) — frontal headache
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
lethargic (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
night sweats (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 1 (1) — runny nose/ sinus congestion/stuffy nose/ nasal congestion/ sneezing/ cough
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) — anemia/low hemoglobin/ low hematocrit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes